CLINICAL TRIAL: NCT02426788
Title: The PRINCE Secondary Study: Persistent Physical Symptoms Reduction Intervention: a System Change and Evaluation in Secondary Care
Brief Title: CBT Plus SMC Compared to SMC for Persistent Physical Symptoms in Secondary Care (PRINCE)
Acronym: PRINCE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King's College London (Other)
Collaborators: South London and Maudsley NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STR130202 (Secondary)
Record Dates: First submitted 2015-04-22; First posted 2015-04-27 (Estimated); Last update posted 2019-05-09 (Actual); Status verified 2018-08

CONDITIONS: Persistent Physical Symptoms (PPS)
Keywords: medically unexplained; fibromyalgia; postural orthostatic tachycardia syndrome (PoTs); non-cardiac chest pain; CFS; irritable bowel syndrome (IBS); functional neurological; chronic pain; hyperventilation; unexplained cough
MeSH Terms: conditions — Fibromyalgia; Postural Orthostatic Tachycardia Syndrome; Irritable Bowel Syndrome; Chronic Pain; Hyperventilation | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- CBT+SMC (Experimental): Cognitive behavioural therapy + Standard Medical Care (cognitive-behavioural therapy+SMC):
  8 hour-long manual-based CBT sessions with a therapist, weekly or fortnightly.
  Interventions: Behavioral: Cognitive behavioural therapy (CBT)
- Standard Medical Care (SMC) (No Intervention): Participants assigned to the SMC group (i.e., control group) will receive all the treatment and support they would otherwise receive outside of a research trial.

INTERVENTIONS:
Behavioral: Cognitive behavioural therapy (CBT) — Behavioral: Cognitive behavioural therapy (CBT) The CBT intervention used in the trial has been adapted for people with PPS and it is based on a model of understanding PPS (Deary et al 2007). The therapy aims to help the patient develop an understanding of the relationship between cognitive, physiological and behavioural aspects of their problem; to understand factors that may be maintaining the problem and to learn how to modify their behavioural and cognitive responses in order to improve quality of life. The approach is transdiagnostic in that it targets processes and underlying mechanisms that affect disorders similarly, rather than focusing on how they are diagnostically different. The approach is personalised during therapy following a detailed assessment.
  Arms: CBT+SMC

SUMMARY:
Brief Summary: Persistent Physical Symptoms (PPS), also known as medically unexplained symptoms (MUS) is a term used to describe a range of persistent bodily symptoms for which the exact cause is unclear. Between 20 and 40% of patients in primary care, and about 50% in secondary care experience PPS. Not only are PPS common, but the overlap across different patient groups may indicate that these phenomena are transdiagnostic. PPS are associated with profound disability and high health care costs, and if left untreated the prognosis of these patients is poor. There is an accumulating body of evidence demonstrating that cognitive behavioural interventions can reduce levels of symptoms and improve functioning in patients with PPS. A pragmatic randomised controlled trial (RCT) was designed to evaluate the clinical and cost-effectiveness of cognitive behavioural therapy (CBT) + Standard Medical Care (SMC) versus Standard Medical Care alone, in the treatment of patients with PPS. The trial will focus on patients with a variety of symptoms (e.g., non-cardiac chest pain, fibromyalgia), across secondary care clinics (e.g., neurology, cardiology, and rheumatology).

DETAILED DESCRIPTION:
Background and study aims In primary care between 20 and 40% of patients have medically unexplained physical symptoms. The term medically unexplained symptoms (MUS) is commonly used by health care professionals. However a survey of a healthy population and a separate survey of patients with chronic fatigue syndrome (CFS) suggested that the term persistent physical symptoms (PPS) was the preferred term. The term PPS may have its drawbacks, but it will be used in the rest of this document to cover MUS as well as any other terms that may be used in the literature and clinical settings to refer to these symptoms. In secondary care, about 50% of patients have PPS, in many specialties. PPS are associated with profound disability and high health care costs. Around 50% of sufferers have co-morbid anxiety and depression and sleep problems. Left untreated, the prognosis of these patients is poor.

This study is a pragmatic RCT that will evaluate the clinical and cost-effectiveness of cognitive behavioural therapy + standard medical care (CBT+SMC), which involves 8 sessions of CBT, versus standard medical care (SMC) in the treatment of patients with PPS.

Who can participate? Patients with various PPS, such as fibromyalgia, non-cardiac chest pain, irritable bowel syndrome and a range of neurological symptoms e.g., weakness will be recruited. Participants will be recruited from clinics in secondary care (e.g., neurology, cardiology, rheumatology) at various hospitals in London.

What does the study involve? Potential participants will be identified by clinical staff who will refer them to the research team. Patients who give their consent to take part in the study will complete a number of questionnaires asking about their symptoms and use of health care services, and about their thoughts, feelings, and beliefs related to their PPS (i.e., baseline). This will take approximately 1.5 hours. After this research assessment, half of participants will be randomly assigned to the treatment arm (CBT+SMC), or to the control (SMC) arm. Participants in the treatment arm will receive 8 individual sessions of CBT (weekly or fortnightly sessions). The therapy aims to help the patient develop an understanding of the relationship between cognitive, physiological and behavioural aspects of their problem; to understand factors that may be maintaining the problem and to learn how to modify their behavioural and cognitive responses in order to improve their quality of life. Participants in the SMC group will receive usual medical care within the clinic.

Participants in both arms will also be asked to complete questionnaires at 9, 20, 40, and 52 weeks after randomisation. The assessment will be independent of the health care professionals delivering care.

What are the possible benefits and risks of participating? By taking part in the study patients may get helpful information about their condition. If assigned to the CBT+SMC arm, patients will receive 8 sessions of CBT focused on helping them manage their symptoms, which may improve their symptoms and increase their psychosocial functioning. It is unclear whether CBT for patients with PPS is effective; this trial will assess whether there are benefits to receiving it. Patients may benefit from being followed up closely and completing measures. It is not expected that participation in the study is associated with risks. The therapists involved in the trial are highly qualified specialists with extensive experience in treating patients with PPS. The trial team also includes a psychiatrist who will further ensure patient safety in complex cases. Participants will be free to take a break at any point during the meetings and are free to withdraw from the study at any point. Participants will also be informed that they can raise any concerns they may have with the research team and will be provided with the Patient Advice & Liaison Service contact information.

Where is the study run from? The study has been set up by the Institute of Psychiatry, Psychology and Neuroscience (IoPPN) at King's College London and the South London and Maudsley National Health Service (NHS) Foundation Trust, and will be conducted at several hospitals in London/Greater London, including Guy's and St Thomas' Hospitals, King's College Hospital, Princess Royal University Hospital, Royal Free Hospital, University Hospital Lewisham and Queen Elizabeth Hospital.

When is the study starting and how long is it expected to run for? The study has started in July 2015 and the end date for the project is March 2019.

Who is funding the study? The study is funded by the Guy's and St. Thomas' Charity.

Who is the main contact? Prof Trudie Chalder trudie.chalder@kcl.ac.uk

ELIGIBILITY:
* Adults (18 - 70 yrs)
* Patients with PPS from broad patient populations (e.g., fibromyalgia, non-cardiac chest pain, postural orthostatic tachycardia syndrome, neurological symptoms);
* Significant functional impairment/moderately severe disability - as indicated by the Work and Social Adjustment Scale (WSAS) score (i.e., a minimum score of 10);
* Ability to complete diaries and questionnaires in English;
* Willingness to complete all trial visits;
* Ability to give written informed consent.

Exclusion Criteria:

* Active psychosis;
* Factitious disorder;
* Headaches as the only PPS;
* Non-epileptic seizures
* Current alcohol dependence or drug addiction as assessed by the clinician;
* Current benzodiazepine use exceeding the equivalent of 10mg diazepam/day;
* The patient is currently receiving CBT/CBT based approach psychotherapy, or has received CBT/CBT based approach psychotherapy in the past year, for their PPS;
* The patient is thought to be at imminent risk of self-harm;
* Patient is taking part in PRINCE Primary trial.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2015-07; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Work and social adjustment scale | 52 weeks post randomisation
  Measures impairment in functioning

SECONDARY OUTCOMES:
Persistent Physical Symptom Questionnaire | 52 weeks post randomisation
  Measures severity, distress, interference and problematic nature of PPS
Patient Health Questionnaire-15 (PHQ-15) | 52 weeks post randomisation
  Measures physical symptoms severity
Patient Health Questionnaire-9 (PHQ-9) | 52 weeks post randomisation
  Measures mood
Generalized Anxiety Disorder-7 (GAD-7) | 52 weeks post randomisation
  Measures generalised anxiety
Clinical Global Impression (CGI) | 52 weeks post randomisation
  Measures patient's perception of their general health improvement
Client Service Receipt Inventory (CSRI) | 52 weeks post randomisation
  Measures health care service receipt, direct and indirect costs of illness, and cost-effectiveness of interventions
EuroQol-5D (EQ-5D) | 52 weeks post randomisation
  Measures health outcome
Cognitive Behavioural Responses Questionnaire | 52 weeks post randomisation
  Measures beliefs and behaviours
Acceptance scale | 52 weeks post randomisation
  assesses degree of acceptance of difficult symptoms

OTHER OUTCOMES:
PSYCHLOPS | 52 weeks post randomisation
  Measures improvement of patient-defined self-rated problems

CONTACTS AND LOCATIONS:
Overall Officials: Trudie Chalder, PhD, Principal Investigator — King's College London
Locations (7):
- United Kingdom (7):
  - Guy's Hospital, London
  - King's College Hospital, London
  - Queen Elizabeth Hospital, London
  - Royal Free Hospital, London
  - St Thomas' Hospital, London
  - University Hospital Lewisham, London
  - Princess Royal University Hospital, Orpington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chalder T, Patel M, James K, Hotopf M, Frank P, Watts K, McCrone P, David A, Ashworth M, Husain M, Garrood T, Moss-Morris R, Landau S. Persistent physical symptoms reduction intervention: a system change and evaluation in secondary care (PRINCE secondary) - a CBT-based transdiagnostic approach: study protocol for a randomised controlled trial. BMC Psychiatry. 2019 Oct 22;19(1):307. doi: 10.1186/s12888-019-2297-y. PMID 31640632